CLINICAL TRIAL: NCT05895110
Title: To Evaluate the Immunogenicity and Safety of Sequentially Enhanced Recombinant Novel Coronavirus Vaccine (CHO Cells) in Patients Aged 3-17 Years After Completion of Two Doses of Novel Coronavirus Inactivated Vaccine
Brief Title: To Evaluate the Immunogenicity and Safety of Sequential Booster Immunization of Recombinant Novel Coronavirus Vaccine (CHO Cells) for SARS-CoV-2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Anhui Zhifei Longcom Biologic Pharmacy Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: LKM-2022-NCV-JQ01
Record Dates: First submitted 2023-05-22; First posted 2023-06-08 (Actual); Last update posted 2023-06-08 (Actual); Status verified 2023-06

CONDITIONS: COVID-19
Keywords: COVID-19 vaccine
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental group (Experimental): 1 dose of the test recombinant novel coronavirus vaccine (CHO cell) was injected into the deltoid muscle of the subject's upper arm
  Interventions: Biological: Recombinant Novel Coronavirus vaccine (CHO Cells)

INTERVENTIONS:
Biological: Recombinant Novel Coronavirus vaccine (CHO Cells) — The experimental vaccine dose used in this study is 25μg/0.5mL. All subjects recruited should have received two doses of novel Coronavirus inactivated vaccine on the market for 6-9 months, and all eligible subjects will receive one dose of recombinant Novel Coronavirus vaccine (CHO cells).

SUMMARY:
An open experimental design was used in this study, and 240 subjects were planned to be enrolled. To evaluate the immunogenicity and safety of recombinant Novel Coronavirus vaccine (CHO cells) after sequential intensification in populations vaccinated with two doses of marketed Novel Coronavirus inactivated vaccine.

DETAILED DESCRIPTION:
One dose of recombinant novel coronavirus vaccine (CHO cell) for test was injected into the upper arm deltoid muscle muscle of the subject

ELIGIBILITY:
Inclusion Criteria:

1. Healthy subjects aged 3 to 17 years who can provide vaccination information proving that they have received two doses of commercially available Novel Coronavirus inactivated vaccine in the last 6-9 months;
2. The subject voluntarily agrees to participate in the study (and/or the subject's legal guardian voluntarily agrees to allow the child to participate in the study), and the guardian and the subject (aged 8-17) sign the informed consent, and can provide valid identification; Understand and comply with test protocol requirements;
3. Armpit temperature < 37.3℃ (> 14 years old), armpit temperature < 37.5℃ (≤14 years old);
4. Female subjects of reproductive age agree to use effective contraceptive measures from the beginning to the end of the study.

Exclusion Criteria:

1. History of confirmed or asymptomatic coronavirus infection or positive nucleic acid test of novel Coronavirus infection;
2. SARS virus disease history or SARS-COV-2 history;
3. Have taken antipyretics or painkillers within 24 hours before vaccination;
4. Have a history of severe allergy to any component of the test vaccine, including aluminum preparation, such as anaphylactic shock, allergic laryngeal edema, allergic purpura, thrombocytopenic purpura, local allergic necrosis reaction (Arthus reaction), dyspnea, angiopantic edema, etc.;
5. Persons suffering from the following diseases:

   1. In the past 7 days, have suffered from digestive diseases (such as diarrhea, abdominal pain, vomiting, etc.);
   2. congenital malformations or developmental disorders, genetic defects, severe malnutrition, etc.;
   3. have thrombocytopenia, any coagulation dysfunction or receive anticoagulant treatment, etc.;
   4. Neurological disorders or neurodysplasia (e.g., migraines, epilepsy, stroke, seizures in the last three years, encephalopathy, focal neurological deficits, Guillain-Barre syndrome, encephalomyelitis or transverse myelitis); History of mental illness or family history;
   5. History of congenital or acquired immune deficiency or autoimmune disease or treatment with immunomodulators within 6 months, such as immunosuppressive doses of glucocorticoids (dose reference: equivalent to prednisone 20mg/ day, over a week); Or monoclonal antibodies; Or thymosin; Or interferon; However, topical use (such as ointments, eye drops, inhalants or nasal sprays) is allowed;
   6. Known to have been diagnosed with an infectious disease, such as active tuberculosis, viral hepatitis or treponema pallidum;
6. Subunit vaccine and inactivated vaccine should be administered within 14 days before experimental vaccine, and live attenuated vaccine should be administered within 30 days before experimental vaccine;
7. Have received blood or blood-related products, including immunoglobulin, within 3 months prior to the trial vaccine; Or planned for use during the study period;
8. People aged 3-17 years who have participated in or are participating in other COVID-19 related clinical trials or have received other COVID-19 vaccines, except those who have completed two doses of marketed Novel Coronavirus inactivated vaccine within 6-9 months;
9. Pregnant (including positive urine pregnancy), or breast-feeding; The Investigator believes that the subject has any disease or condition that may place the subject at unacceptable risk; Subjects cannot meet the requirements of the program; Conditions that interfere with the assessment of vaccine response.

Ages: 3 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 240 (Actual)
Dates: Start 2022-04-29 (Actual); Primary Completion 2022-11-19 (Actual); Study Completion 2022-11-19 (Actual)

PRIMARY OUTCOMES:
SARS-COV-2 neutralizing antibody | 14 days and 6 months after inoculation
  Titers of SARS-COV-2 neutralizing Antibody at 14 days and 6 months after vaccination of recombinant Novel Coronavirus vaccine (CHO cells) (GMT)

SECONDARY OUTCOMES:
SARS-COV-2 neutralizing antibody | 14 days and 6 months after inoculation
  GMI and 4-fold increase in SARS-COV-2 neutralizing antibody at 14 days and 6 months after intensification of recombinant Novel Coronavirus vaccine (CHO cells)

CONTACTS AND LOCATIONS:
Locations (1):
- Hunan Provincial Center for Disease Control and Prevention, Changsha, Hunan, China

REFERENCES:
- [Derived] Huang T, Hu Q, Zhou X, Yang H, Xia W, Cao F, Deng M, Teng X, Ding F, Zhong Z, Gao L, Sun J, Gong L. Immunogenicity and safety of a recombinant COVID-19 vaccine (ZF2001) as heterologous booster after priming with inactivated vaccine in healthy children and adolescents aged 3-17 years: an open-labeled, single-arm clinical trial. BMC Infect Dis. 2024 Apr 19;24(1):413. doi: 10.1186/s12879-024-09293-1. PMID 38641791